CLINICAL TRIAL: NCT02417987
Title: High Volume Injection (HVI) or Autologous Conditioned Plasma (ACP) in Chronic Achilles Tendinopathy: A Randomized Controlled Double Blinded Trial
Brief Title: High Volume Injection or Autologous Conditioned Plasma (ACP) in Chronic Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Anders Ploug Boesen, MD, PhD., Bispebjerg Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: H-1-2010-052a
Record Dates: First submitted 2014-11-04; First posted 2015-04-16 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Tendinopathy
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Volume injection (Active Comparator): A total volume of 50 ml:
  * 10 mls 0.5% bupivacaine hydrochloride and
  * 20 mg of Depomedrol (hydrocortisone)
  * 40 mls saline (NaCl) HVI is injected one time at baseline and thereafter the group received sham treatment at 2 weeks, 4 weeks and after 6 weeks.
  Interventions: Other: Placebo; Biological: Autologous conditioned plasma (ACP)
- Autologous conditioned plasma (ACP) (Active Comparator): Whole blood was drawn from the patients using arthrex system (total of 10 mls whole blood). After that the whole blood is spined for 5 minutes and ACP with platelets and growth factors is separated from the red and white blood cells (4 mls).
  The ACP is injected 4 times (at baseline, 2 weeks, 4 weeks and after 6 weeks)
  Interventions: Other: Placebo; Drug: High Volume injection
- Placebo (Sham Comparator): A few drops of saline is injected in the soft tissue away from the tendon.
  Interventions: Drug: High Volume injection; Biological: Autologous conditioned plasma (ACP)

INTERVENTIONS:
Other: Placebo — The skin was penetrated with a needle and few drops of saline injected in the soft tissue away from the tendon
  Other Names: Sham treatment
  Arms: Autologous conditioned plasma (ACP); High Volume injection
Drug: High Volume injection — Injection with10 mls 0.5% bupivacaine hydrochloride and 20 mg of Depomedrol 40 mls saline (NaCl) around the tendon
  Other Names: HVI
  Arms: Autologous conditioned plasma (ACP); Placebo
Biological: Autologous conditioned plasma (ACP) — Injection with 4 mls of ACP around the tendon
  Other Names: Platelet-rich plasma (PRP)
  Arms: High Volume injection; Placebo

SUMMARY:
The aim of the study is to examine patients with chronic Achilles Tendinopathy (AT) and to compare the effect of high volume injection (HVI) or autologous conditioned plasma (ACP) in combination with eccentric training to placebo treatment (sham treatment combined with eccentric exercises).

Healthy males with AT will be randomly assigned to either 1) HVI (50 mls;10 mls 0.5% bupivacaine hydrochloride and 20 mg of Depomedrol followed by 40 mls saline), 2) ACP (~ 4 mls) or 3) Placebo (Plc) treatment. All subjects will perform a 12-wk eccentric training program and examinations will be done at baseline (before treatment) with follow-ups after 6 weeks, 12 weeks and again after 24 weeks prior to baseline to see any possible changes and differences between groups (HVI, ACP and Plc)

DETAILED DESCRIPTION:
Chronic Achilles tendinopathy (AT) is a common and impairing disorder. Only sparse scientific evidence exists for the present used treatments and no golden standard treatment exists so far.

Aim: The aim of the study is in AT patients to examine and compare the effect of high volume injection (HVI) or autologous conditioned plasma (ACP) in combination with eccentric training to placebo treatment (sham treatment and eccentric exercises).

Materials and methods: Healthy males (21-59 years; n=60) with AT is randomly assigned to either 1) HVI (50 mls;10 mls 0.5% bupivacaine hydrochloride and 20 mg of Depomedrol followed by 40 mls saline), 2) ACP (~ 4 mls) or 3) placebo (Plc) treatment. Participants will treated on 4 successive occasions with 2 weeks (wks) interval (HVI will only be injected once at baseline, the 3 following injections will be placebo). The injections will be performed under ultrasound guidance. All subjects will undergo a 12-wk eccentric training program. Clinical effects will be assessed as changes in symptoms and pain (VISA-A and VAS score), tendon ultrasound thickness and muscle function (one-legged heel-rise test). All outcome measures will be recorded at baseline and again at 6 weeks, 12 week and 6 month follow-up.

Results: Will se the changes and differences between groups (HVI, ACP and Placebo) in VISA-A scores, VAS scores, ultrasound (tendon thickness) and muscle function.

Statistics: All data will be analyzed in SigmaPlot v11 using two-way repeated measures ANOVA with Student-Newman-Keuls Post-hoc test. This is used to see changes over time in all groups (time effect) and differences between groups within time-points (group effect). All data will be presented as mean ± SEM time.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and ultrasound diagnosed unilateral midt-tendinous achilles tendinopathy
* Symptoms > 3 month
* No steroid injections < 6 month
* 60 males with BMI <30 between 18-60 years.

Exclusion Criteria:

* Bilateral achilles tendinopathy
* Insertional tendinopathy
* Steroid injections < 6 month
* Diabetes or cardiovascular disease
* Smoking
* Treatment with fluoroquinolones < 6 month

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
VISA-A score | Baseline, 6 weeks, 12 weeks and 24 weeks
  See the changes in VISA-A score over time due to the effect of treatment between groups (HVI, ACP and Plc)

SECONDARY OUTCOMES:
VAS score | Baseline, 6 weeks, 12 weeks and 24 weeks
  See the changes in VAS score over time due to the effect of treatment between groups (HVI, ACP and Plc)
Ultrasound tendon thickness and doppler activity | Baseline, 6 weeks, 12 weeks and 24 weeks
  See the changes in tendon thickness over time due to the effect of treatment between groups (HVI, ACP and Plc)

OTHER OUTCOMES:
Muscle function performance test (total workload) | Baseline, 6 weeks, 12 weeks and 24 weeks
  See the muscle function performance (total workload- heel raise test) performed over time due to the effect of treatment between groups (HVI, ACP and Plc)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjaer, Dr. Med., Principal Investigator — Institute of Sportsmedicine Copenhagen, Bispebjerg Hospital

REFERENCES:
- [Derived] Boesen AP, Hansen R, Boesen MI, Malliaras P, Langberg H. Effect of High-Volume Injection, Platelet-Rich Plasma, and Sham Treatment in Chronic Midportion Achilles Tendinopathy: A Randomized Double-Blinded Prospective Study. Am J Sports Med. 2017 Jul;45(9):2034-2043. doi: 10.1177/0363546517702862. Epub 2017 May 22. PMID 28530451